CLINICAL TRIAL: NCT05024409
Title: Use of Low Cost Orthotic Device to Improve Upper Extremity Function in Children With Cerebral Palsy
Brief Title: Cerebral Palsy Upper Extremity Orthotic Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Alice Chu, MD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2020000653
Record Dates: First submitted 2021-08-03; First posted 2021-08-27 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthotic + Occupational Therapy (Experimental)
  Interventions: Device: Upper Extremity Orthotic
- Occupational Therapy alone (Active Comparator)
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Device: Upper Extremity Orthotic — 3D printed orthotic which uses elbow motion to facilitate finger extension
  Arms: Orthotic + Occupational Therapy
Other: Occupational Therapy — 6 weekly sessions of occupational therapy, without use of an assistive orthotic device
  Arms: Occupational Therapy alone

SUMMARY:
Upper extremity therapies for children with cerebral palsy (CP) have been validated for improving function in higher functioning patients. Those who function at the lowest end of the scale, on the Manual Ability Classification System scale (MACS) III-V, comprise 34-54% of the population, but as yet have no evidence-based interventions specific to their needs. Lower functioning children often retain some voluntary control of the elbow in spite of limited finger motion. A dynamic splint, or exoskeleton, could utilize the tenodesis effect from elbow motion to drive finger release while retaining flexor tone for grasp, potentially creating a portable, home-based therapeutic tool. The purpose of this study is to assess the effectiveness of an upper extremity orthotic device in improving the upper extremity function of children with cerebral palsy who have limited use of their hands.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cerebral palsy, age 4-17 years, moderate-severe hand disability as graded by the Manual Ability Classification System, active movement of the elbow, ability to follow commands and participate in goal-making and repetitive tasks

Exclusion Criteria:

* mild or extremely severe hand disability, Botox or orthopaedic surgery within the past 6 months, severe contractures, lack of voluntary arm motion, unable to follow commands due to severe cognitive impairment

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment from 1) pre to post treatment; 2) post treatment to 3 month followup, and 3) pre treatment to 3 mos after cessation of treatment | through study completion, an average of 6 months
  The Assisting Hand Assessment (AHA) is a test of hand function in children with difficulties using one of their hands. The AHA measures how effectively the affected hand and arm is used in bimanual performance. An assessment is performed by observing the child's spontaneous handling of toys in a relaxed and playful session. The scale is 0-100, and a higher score indicates better function. A change of +5 is clinically significant.
Change in Melbourne Assessment-2 from 1) pre to post treatment; 2) post treatment to 3 month followup, and 3) pre treatment to 3 mos after cessation of treatment | through study completion, an average of 6 months
  The Melbourne Assessment 2 (MA2) is a valid and reliable criterion-referenced test for evaluating four elements of upper limb movement quality in children with a neurological impairment aged 2.5 to 15 years: (i) Range of movement, (ii) Accuracy of reach and placement, (iii) Dexterity of grasp, release and manipulation and (iv) Fluency of movement.
  The full test comprises 14 test items which require a child to reach to, grasp, release and manipulate simple objects. Each child's test performance is video recorded for subsequent scoring.
  Scoring is completed across the 30 score items using a three, four or five point scale and individually defined scoring criteria. Item scores relating to each element of movement measured are summed within the corresponding sub-scale. A raw score scale change of 3 for range of motion, dexterity, and fluency; and a change of 4 for accuracy is considered clinically significant.
Change in Children's Hand Use Experience Questionnaire from 1) pre to post treatment; 2) post treatment to 3 month followup, and 3) pre treatment to 3 mos after cessation of treatment | through study completion, an average of 6 months
  CHEQ is a newly developed questionnaire. It has been developed for children and adolescents with decreased function in one hand, for example hemiplegic CP, obstetric brachial plexus palsy (OBPP) and upper limb reduction deficiency, and for their parents. The scale is 0-100, with the higher score indicating better abilities.
Change in range of motion for shoulder, elbow, forearm, wrist, and fingers from 1) pre to post treatment; 2) post treatment to 3 month followup, and 3) pre treatment to 3 mos after cessation of treatment | pre treatment, immediate post treatment, and 3 month followup

SECONDARY OUTCOMES:
Change in motion analysis parameters from 1) pre to post treatment; 2) post treatment to 3 month followup, and 3) pre treatment to 3 mos after cessation of treatment | pre treatment, immediate post treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rutgers NJMS, Newark, New Jersey
  - Children's Specialized Hospital, Union, New Jersey

IPD SHARING:
Plan to Share IPD: No